CLINICAL TRIAL: NCT00197743
Title: Trial of Vitamins in HIV Progression and Transmission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Wafaie Fawzi, Harvard School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD32257
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: HIV Infections; Disease Transmission, Vertical
Keywords: HIV; Multivitamins; Pregnancy outcomes; Tanzania; Women
MeSH Terms: conditions — HIV Infections | interventions — Vitamin A; beta Carotene; Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin A (Active Comparator): Vitamin A + Beta Carotene
  Interventions: Dietary Supplement: Vitamin A + Beta Carotene
- Multivitamins (Active Comparator): Vitamins B, C, and E
  Interventions: Dietary Supplement: Multivitamins
- Vitamin A + Multivitamins (Active Comparator): Vitamin A + Beta Carotene, Vitamins B, C, and E
  Interventions: Dietary Supplement: Vitamin A + Beta Carotene; Dietary Supplement: Multivitamins
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin A + Beta Carotene — one daily oral dose of 30 mg beta-carotene + 5000 IU preformed vitamin A
  Arms: Vitamin A; Vitamin A + Multivitamins
Dietary Supplement: Multivitamins — one daily oral dose of 20 mg thiamine (vitamin B-1), 20 mg riboflavin (vitamin B-2), 25 mg vitamin B-6, 100 mg niacin, 50 ug cobalamin (vitamin B-12), 500 mg vitamin C, 30 mg vitamin E, and 0.8 mg folic acid
  Arms: Multivitamins; Vitamin A + Multivitamins
Other: Placebo — Placebo pill
  Arms: Placebo

SUMMARY:
This study tested the hypothesis that multivitamin supplementation given to HIV+ pregnant women in Tanzania would slow disease progression and enhance their overall health.

DETAILED DESCRIPTION:
In this study, we sought to examine whether the administration of multivitamins excluding vitamin A, multivitamins including vitamin A, or vitamin A alone would reduce the risk of perinatal transmission of HIV and slow the rate of disease progression in a group of pregnant HIV infected women. We also examined the efficacy of the supplements on pregnancy outcomes, and risks of maternal and child morbidity and wasting.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected women presenting to antenatal care between 12 and 27 weeks of gestation:

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1085 (Actual)
Dates: Start 1995-04; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
To examine the effect of multivitamin and/or Vitamin A supplements on the risk of perinatal transmission of HIV and rate of HIV disease progression | until the end of follow-up in August, 2003

SECONDARY OUTCOMES:
To examine the effect of multivitamin and/or Vitamin A supplements on child and maternal morbidity, child growth and child mortality | until the end of follow-up in August 2003

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MD,DrPh, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard School of Public Health, Boston, Massachusetts, United States

REFERENCES:
- [Result] Fawzi WW, Msamanga GI, Spiegelman D, Wei R, Kapiga S, Villamor E, Mwakagile D, Mugusi F, Hertzmark E, Essex M, Hunter DJ. A randomized trial of multivitamin supplements and HIV disease progression and mortality. N Engl J Med. 2004 Jul 1;351(1):23-32. doi: 10.1056/NEJMoa040541. PMID 15229304
- [Result] Fawzi WW, Msamanga GI, Hunter D, Renjifo B, Antelman G, Bang H, Manji K, Kapiga S, Mwakagile D, Essex M, Spiegelman D. Randomized trial of vitamin supplements in relation to transmission of HIV-1 through breastfeeding and early child mortality. AIDS. 2002 Sep 27;16(14):1935-44. doi: 10.1097/00002030-200209270-00011. PMID 12351954
- [Result] Fawzi WW, Msamanga G, Hunter D, Urassa E, Renjifo B, Mwakagile D, Hertzmark E, Coley J, Garland M, Kapiga S, Antelman G, Essex M, Spiegelman D. Randomized trial of vitamin supplements in relation to vertical transmission of HIV-1 in Tanzania. J Acquir Immune Defic Syndr. 2000 Mar 1;23(3):246-54. doi: 10.1097/00126334-200003010-00006. PMID 10839660
- [Result] Fawzi WW, Msamanga GI, Spiegelman D, Urassa EJ, McGrath N, Mwakagile D, Antelman G, Mbise R, Herrera G, Kapiga S, Willett W, Hunter DJ. Randomised trial of effects of vitamin supplements on pregnancy outcomes and T cell counts in HIV-1-infected women in Tanzania. Lancet. 1998 May 16;351(9114):1477-82. doi: 10.1016/s0140-6736(98)04197-x. PMID 9605804
- [Derived] Khavari N, Jiang H, Manji K, Msamanga G, Spiegelman D, Fawzi W, Duggan C. Maternal multivitamin supplementation reduces the risk of diarrhoea among HIV-exposed children through age 5 years. Int Health. 2014 Dec;6(4):298-305. doi: 10.1093/inthealth/ihu061. Epub 2014 Aug 30. PMID 25173342
- [Derived] Natchu UC, Liu E, Duggan C, Msamanga G, Peterson K, Aboud S, Spiegelman D, Fawzi WW. Exclusive breastfeeding reduces risk of mortality in infants up to 6 mo of age born to HIV-positive Tanzanian women. Am J Clin Nutr. 2012 Nov;96(5):1071-8. doi: 10.3945/ajcn.111.024356. Epub 2012 Oct 10. PMID 23053555